CLINICAL TRIAL: NCT01271920
Title: A Phase Ib/II, Multi-center, Open-label Study to Evaluate the Efficacy of AUY922 in Combination With Trastuzumab in Patients With Locally Advanced or Metastatic HER2-positive Breast Cancer, That Has Progressed After or During at Least One Trastuzumab-containing Regimen
Brief Title: Combination of AUY922 With Trastuzumab in HER2+ Advanced Breast Cancer Patients Previously Treated With Trastuzumab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAUY922A2109; 2009-015628-27 (EudraCT Number)
Record Dates: First submitted 2010-11-03; First posted 2011-01-07 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2017-02

CONDITIONS: Advanced HER2-positive Breast Cancer
Keywords: Trastuzumab-refractory; advanced HER2-positive breast cancer,; Hsp90,; 2nd or 3rd line treatment
MeSH Terms: conditions — Neoplasm Metastasis | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide; Trastuzumab

ARMS (1):
- AUY922 + Trastuzumab (Experimental)
  Interventions: Drug: AUY922; Drug: Trastuzumab

INTERVENTIONS:
Drug: AUY922
Drug: Trastuzumab

SUMMARY:
The phase Ib part of the trial will assess the MTD of AUY922 in combination with Trastuzumab in patients with Trastuzumab-refractory locally advanced or metastatic HER2+. The MTD is defined as the highest drug dosage not causing in the first cycle of treatment (28 days) medically unacceptable dose limiting toxicity (DLT).

The phase II part of the trial will assess any potential effect on efficacy of adding AUY922 to Trastuzumab in patients with Trastuzumab-refractory locally advanced or metastatic HER2+ breast cancer.

Both AUY922 and Trastuzumab will be administered as a weekly IV infusion. Treatment should be continued as long as the patient does not have disease progression and tolerates the treatment. The following reasons are examples of acceptable reasons for discontinuing the study; tumor progression (by RECIST, as assessed by the investigator), unacceptable toxicity, death, or discontinuation from the study for any other reason, such as patient refusal, withdrawn consent, lost to follow-up or investigator decision.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with confirmed HER-2 positive , non-operable locally advanced or metastatic breast cancer
* All patients must have received at least 1 but no more than 2 prior anti HER2 based regimens including at least 1 regimen containing Trastuzumab.
* All patients must have at least one measurable lesion as defined by RECIST criteria.
* All patients must have documented progressive disease following the last line of therapy before entering the study
* ECOG Performance status ≤ 1

Exclusion Criteria:

* Patients with known CNS metastasis which are: symptomatic or require treatment for symptom control and/or growing
* Prior treatment with any HSP90 or HDAC inhibitor
* Impaired cardiac function
* Acute or chronic liver or renal disease
* Patients who are currently receiving treatment with any medication which has a relative risk of prolonging the QTc interval or inducing Torsades de Pointes and cannot be switched or discontinued to an alternative drug prior to commencing AUY922
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
* Patients who do not have either an archival tumor sample available or are unwilling to have a fresh tumor sample collected at baseline.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and/or recommended phase two dose (RPTD) of AUY922 in combination with Trastuzumab (phase lb) | 4 weeks
Overall Response Rate as assessed by RECIST (phase ll) | Every 8 weeks for the first 24 weeks and every 12 weeks thereafter

SECONDARY OUTCOMES:
Assess concentration of AUY922 and BJP762 in the blood at different time points (phase lb & ll) | 4 weeks
Assess frequency, intensity and duration of Adverse Events as a Measure of Safety and Tolerability (phase lb & ll) | average 6 months
Progression Free Survival (PFS) at the RPTD dose (phase ll only) | every 3 months until 24 months after the last patient has been enrolled
Overall Survival (OS) at the RPTD dose | every 3 months until 24 months after the last patient has been enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Investigative Site, Study Director — Novartis Investigative Site
Locations (16):
- Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas, United States
- France (2):
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Saint-Herblain Cédex
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Tübingen
- Italy (2):
  - Novartis Investigative Site, Prato, PO
  - Novartis Investigative Site, Candiolo, TO
- Novartis Investigative Site, Singapore, Singapore
- Spain (3):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Stockholm, Sweden
- United Kingdom (4):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Oxford

REFERENCES:
- [Result] Kong A, Rea D, Ahmed S, Beck JT, Lopez Lopez R, Biganzoli L, Armstrong AC, Aglietta M, Alba E, Campone M, Hsu Schmitz SF, Lefebvre C, Akimov M, Lee SC. Phase 1B/2 study of the HSP90 inhibitor AUY922 plus trastuzumab in metastatic HER2-positive breast cancer patients who have progressed on trastuzumab-based regimen. Oncotarget. 2016 Jun 21;7(25):37680-37692. doi: 10.18632/oncotarget.8974. PMID 27129177
- See also: Results for CAUY922A2109 can be found on the Novartis Clinical Trials Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12663